CLINICAL TRIAL: NCT06394323
Title: UNCPM 22323 - Supporting Oral Pre-exposure Prophylaxis Decision Making Among Pregnant Women in Lilongwe, Malawi: a Pilot Study
Brief Title: Supporting Oral Pre-exposure Prophylaxis Decision Making Among Pregnant Women in Lilongwe, Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-3102; K01MH121186 (NIH)
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: HIV Prevention
Keywords: PrEP in pregnancy and breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- My Choice for HIV Prevention (MyChoice) (Experimental): The MyChoice intervention consists of PrEP shared decision-making counseling delivered by a trained counselor. It begins with a review of HIV risk in pregnancy/breastfeeding including discussion of population-specific risk factors which may apply to the participant. Next, the counselor presents HIV prevention options including daily oral PrEP and internal and external condoms (discussing attributes and potential advantages and disadvantages of each method). This is followed by a values clarification exercise to identify which features of the competing options matter most to the participant (product attributes and personal and interpersonal implications of each method). The counselor reviews information about these valued features for each offered method. This information and checks to understand and address any unmet participant decision support needs serve as the basis for structured deliberation to collaboratively identify participant preferred method(s).
  Interventions: Behavioral: Behavioral: My Choice for HIV Prevention (MyChoice)
- Standard of care (control arm) (Active Comparator): Participants randomized to the control arm will receive PrEP counseling as based on the current standard of care (SOC). The SOC counseling will be delivered by a trained study staff member. The SOC counselor PrEP counseling according to national guidelines. Control arm participants will receive comprehensive education on both the advantages and limitations of oral PrEP, including guidance on potential side effects. The SOC counselor will assess the woman's eligibility, willingness, and readiness to start using PrEP.
  Interventions: Behavioral: Behavioral: My Choice for HIV Prevention (MyChoice)
- Male Partner In-Depth Interviews (No Intervention): Male partners of a subset of women enrolled in the study completed qualitative in-depth interviews. Each male partner completed a single in-depth interview conducted by a trained interviewer using a semi-structured interview guide including topics related to their involvement in the woman's PrEP decision making, attitudes towards women's use of PrEP, role supporting women's use of PrEP, and impact of women's use of PrEP on their use of antiretroviral therapy (if applicable).
- Clinician and Counselor In-Depth Interviews (No Intervention): Study staff including intervention counselors and clinicians completed qualitative in-depth interviews. Each staff member completed a single in-depth interview conducted by a trained interviewer using a semi-structured interview guide including topics related to their impressions of the study counseling, perceptions of participants' decision making regarding PrEP use, opinions regarding future implementation of the study intervention, and experiences with study procedures.

INTERVENTIONS:
Behavioral: Behavioral: My Choice for HIV Prevention (MyChoice) — My Choice for HIV Prevention (MyChoice), is a counselor-delivered shared decision-making approach for pregnant women considering PrEP
  Arms: My Choice for HIV Prevention (MyChoice); Standard of care (control arm)

SUMMARY:
Purpose: The overall objective of this pilot study is to evaluate the feasibility, acceptability, and appropriateness of a shared decision-making (SDM) intervention to support personally appropriate decision making about PrEP use during pregnancy and breastfeeding.

Participants: The primary population to be recruited for this study is HIV-negative pregnant women. For qualitative data collection only, investigators will also recruit male partners of these participants, and PrEP counselors and health care workers. 100 HIV-negative pregnant women will be recruited to participate in the pilot study. A subset of these participants will participate in qualitative interviews. Up to 20 male partners and up to 15 study staff will be recruited to participate in qualitative in-depth interviews.

Procedures (methods): 100 women will be randomized to receive either the SDM intervention addressing daily oral PrEP and alternative HIV prevention methods (condoms), or standard of care counselling addressing the same prevention methods. Investigators will evaluate the feasibility, acceptability, and appropriateness of the intervention and associated study procedures. Women expressing interest in oral PrEP will be referred to government PrEP services.

DETAILED DESCRIPTION:
Study design:

This is a pilot feasibility study of a shared decision making (SDM) intervention for pregnant women considering PrEP. 100 women will be randomized to receive either the SDM intervention addressing daily oral PrEP and alternative HIV prevention methods (condoms), or standard of care counselling addressing the same prevention methods. Investigators will evaluate the feasibility, acceptability, and appropriateness of the intervention and associated study procedures. Women expressing interest in oral PrEP will be referred to government PrEP services.

Study intervention (intervention arm):

The study intervention, My Choice for HIV Prevention (MyChoice), is a counselor-delivered shared decision-making approach for pregnant women considering PrEP. The intervention counseling will be delivered by trained study staff with a background in psychosocial counseling. The intervention consists of counseling facilitated by a SDM tool. The woman's partner may be present depending on her preference. It begins with a review of HIV risk in pregnancy/breastfeeding including discussion of population-specific risk factors which may apply to the participant. After understanding participant HIV risk and desire for HIV protection, the counselor presents HIV prevention options including oral PrEP, and internal and external condoms (discussing attributes and potential advantages and disadvantages of each method). This is followed by a values clarification exercise to identify which features of the competing options matter most to the participant (product attributes and personal and interpersonal implications of each method). The counselor reviews information about these valued features for each offered method. This information and checks to understand and address any unmet participant decision support needs serve as the basis for structured deliberation to collaboratively identify participant preferred method(s). The participant may defer or decline the decision and may request a follow-up counseling visit to take more time to consider her preference or return with a partner or other supporter. If and when a decision is made, the counselor provides post-decision counseling including adherence counseling and disclosure counseling if desired.

Standard of care (control arm):

Participants randomized to the control arm will PrEP counseling as based on the current standard of care (SOC). The SOC counseling will be delivered by a trained study staff member. The SOC counselor PrEP counseling according to national guidelines.Per current guidelines, the SOC counseling may include the following elements: An HIV risk assessment according to PrEP eligibility criteria; discussion of a combination prevention approach (PrEP and condoms) and risk reduction strategies. The women will receive comprehensive education on both the advantages and limitations of PrEP, including guidance on managing potential side effects. Subsequently, the counselor will assess the woman's eligibility, willingness, and readiness to start using PrEP.

Participants choosing oral PrEP during the counselling session in either intervention or comparison arm will receive an assisted referral to government PrEP services at the study site to initiate their selected PrEP method per national guidelines. Initiation of oral PrEP (i.e., receipt of prescription) will be confirmed through clinic or pharmacy records, as well as information on reasons for non-initiation if applicable.

Follow-up:

Participants will complete follow-up visits at month 1, month 2, and month 3. Study visits will be scheduled to align with antenatal care (ANC)/pharmacy visits whenever possible to minimize the number of trips needed at the clinic.

Interviewer-administered questionnaires will be completed at the month 1 and month 3 follow-up visits. Questionnaires will assess study outcomes and associated social and behavioural measures to contextualize understanding of primary study outcomes. A subset of participants will complete in-depth qualitative interviews at month 1. Interviews will provide additional understanding of participant experiences with the intervention and experience using PrEP (if applicable).

At each follow-up visit, women who have chosen oral PrEP will undergo adherence assessment through self-report and pill counts. Furthermore, investigators will collect dried blood spots (DBS) at month 2 to assess adherence among all oral PrEP users (see below).

Biological specimen collection and testing:

To assess quantify drug concentrations to assess PrEP adherence among participants taking up oral PrEP, a participant blood specimen will be collected via venipuncture at the for applicable participants (those using oral PrEP). This specimen will be used to create a dried blood spot (DBS) specimen at the local designated laboratory, prior to storage and shipment to the reference pharmacology laboratory for testing.

All samples will be obtained from study participants by trained study staff according to approved standard operating procedures. All samples will be processed according to the assay manufacturers' specifications. Specimens will be transported, processed, and temporarily housed at UNC Project Malawi (UNCPM) (Lilongwe, Malawi) and shipped to University of North Carolina (UNC) Chapel Hill for analysis. All laboratory testing will be performed by trained staff using standard operating procedures and according to specific assay manufacturers' specifications.

ELIGIBILITY:
The criteria for pregnant women participants is as follows:

Inclusion Criteria:

* Age 18 or older
* Documented pregnancy by urine pregnancy test or physical exam
* Documented negative HIV status within the past three months
* Identified factor(s) for elevated risk for HIV acquisition per PrEP national eligibility guidelines
* Willingness to remain in the study site's catchment area over the course of study follow-up and to comply with visit schedule
* Ability and willingness to provide informed consent

Exclusion Criteria:

* Positive HIV test at time of screening
* No identified HIV risk factors per national PrEP guidelines
* Risk for intimate partner violence or social harms as a result of participation, in the judgement of the study personnel

Investigators will also conduct interviews with male partners and study staff to assess exploratory qualitative outcomes. All study staff will be eligible to participate in an interview. Male partners will be eligible to participate if they meet the following criteria:

* Referred by a study participant as her romantic partner
* Age 18 or older
* Able and willing to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Hill, PhD, MSPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Bwaila Hospital, Lilongwe, Central Region, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Saidi F, Welch S, Phanga T, Sulpizio C, Paile L, Ngo'ma D, Tsidya M, Chindebvu M, Nkhoma G, Nkhalamba L, Kaliati I, Mkochi N, Chakala H, Kumwenda W, Bula A, Winner P, Munthali T, Nyamaizi A, Keys J, Maman S, Pearce L, Golin C, Chi BH, Hill LM. Supporting Oral and Long-Acting HIV Preexposure Prophylaxis Decision-Making Among Pregnant Women (MyChoice Intervention): Protocol for 2 Pilot Randomized Controlled Trials. JMIR Res Protoc. 2025 Nov 13;14:e76442. doi: 10.2196/76442. PMID 41232107

RESULTS

PARTICIPANT FLOW:
Groups:
- My Choice for HIV Prevention (MyChoice): The MyChoice intervention consists of pre-exposure prophylaxis (PrEP) shared decision-making counseling delivered by a trained counselor, administered at month 0 following randomization to this arm. The MyChoice intervention begins with a review of HIV risk in pregnancy and the postpartum period including discussion of population-specific risk factors which may apply to the participant. Next, the counselor presents HIV prevention options including daily oral PrEP and internal and external condoms (discussing attributes and potential advantages and disadvantages of each method). This is followed by a values clarification exercise to identify which features of the competing options matter most to the participant (including product attributes and personal and interpersonal implications of each method). The counselor reviews information about the participant's valued features for each method offered. This information and checks to understand and address any unmet participant decision support needs serve as the basis for structured deliberation to collaboratively identify participant preferred method(s).
- Standard of Care (SOC) Control Arm: Participants randomized to the control arm receive pre-exposure prophylaxis (PrEP) counseling based on the current standard of care (SOC) at month 0 after randomization to this arm. The SOC counseling is delivered by a trained study staff member. The SOC counselor delivers PrEP counseling according to national guidelines. Control arm participants receive comprehensive education on both the advantages and limitations of oral PrEP, including guidance on potential side effects. The SOC counselor assesses each participant's eligibility, willingness, and readiness to start using daily oral PrEP.
Period: Overall Study
Arm/Group | My Choice for HIV Prevention (MyChoice) | Standard of Care (SOC) Control Arm | Male Partner In-Depth Interviews | Clinician and Counselor In-Depth Interviews
Started | 50 | 50 | 20 (Provided informed consent, no primary or secondary outcomes were reported) | 12 (Provided informed consent, no primary or secondary outcomes were reported)
Month 2 | 46 | 42 | 20 | 12
Completed | 46 | 43 | 20 | 12
Not Completed | 4 | 7 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants at baseline who were consented and enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | My Choice for HIV Prevention (MyChoice) | Standard of Care (SOC) Control Arm | Male Partner In-Depth Interviews | Clinician and Counselor In-Depth Interviews | Total
Number analyzed (Participants) | 50 | 50 | 20 | 12 | 132
Age, Categorical [Count of Participants; unit: Participants] — Population: Specific age data were collected for all Arms except the Male Partners but based on Inclusion criteria and counselor interactions, all Male Partners were >/= 18 and </= 65 years of age.
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 50 | 50 | 20 | 12 | 132
    >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Age was not collected for Male Partners.
  years
    number analyzed (Participants) | 50 | 50 | 0 | 12 | 112
    (all) | 24 [22 to 27] | 24 [21 to 28] |  | 35 [27 to 42] | 24 [21 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 0 | 12 | 112
  Male | 0 | 0 | 20 | 0 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 50 | 50 | 20 | 12 | 132
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 50 | 50 | 20 | 12 | 132
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Malawi | 50 | 50 | 20 | 12 | 132

OUTCOME MEASURES:

1. Primary Outcome: Mean Acceptability of Intervention (AIM) Scale Score
Description: Intervention acceptability was defined as the extent to which participants perceived the intervention to be agreeable, palatable, or satisfactory. Acceptability was assessed through participant self-report using a validated 4-item scale (AIM). This scale measures how agreeable and satisfactory women find the intervention (responses rated on a 5-point Likert scale ranging from 1="Completely Disagree" to 5="Completely Agree"). For each participant at each timepoint, a mean AIM scale score was calculated ranging from 1 to 5. Higher scores indicate greater acceptability. Individuals' mean AIM scale scores were averaged at each timepoint, and a 95% confidence interval around the mean of means was calculated using the common standard error.
Time Frame: enrollment visit (month 0), month 2 follow up visit
Population: Only participants that received the MyChoice intervention and had one or more completed items of the AIM scale were included. Participants in the Standard of Care (SOC) Control Arm, Male Partner In-Depth Interviews, and Clinician and Counselor In-Depth Interviews were not asked to complete these items.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- My Choice for HIV Prevention (MyChoice): The MyChoice intervention consists of pre-exposure prophylaxis (PrEP) shared decision-making counseling delivered by a trained counselor, administered at month 0 following randomization to this arm. The MyChoice intervention begins with a review of HIV risk in pregnancy/breastfeeding including discussion of population-specific risk factors which may apply to the participant. Next, the counselor presents HIV prevention options including daily oral PrEP and internal and external condoms (discussing attributes and potential advantages and disadvantages of each method). This is followed by a values clarification exercise to identify which features of the competing options matter most to the participant (product attributes and personal and interpersonal implications of each method). The counselor reviews information about these valued features for each offered method. This information and checks to understand and address any unmet participant decision support needs serve as the basis for structured deliberation to collaboratively identify participant preferred method(s).
- Standard of Care (SOC) Control Arm: Participants randomized to the control arm will receive pre-exposure prophylaxis (PrEP) counseling based on the current standard of care (SOC) at month 0 after randomization to this arm. The SOC counseling will be delivered by a trained study staff member. The SOC counselor delivers PrEP counseling according to national guidelines. Control arm participants will receive comprehensive education on both the advantages and limitations of oral PrEP, including guidance on potential side effects. The SOC counselor will assess the woman's eligibility, willingness, and readiness to start using daily oral PrEP.
Arm/Group | My Choice for HIV Prevention (MyChoice) | Standard of Care (SOC) Control Arm | Male Partner In-Depth Interviews | Clinician and Counselor In-Depth Interviews
Number analyzed (Participants) | 50 | 0 | 0 | 0
score on a scale
  Enrollment (Month 0) | 4.65 [4.52 to 4.77] |  |  |
  Month 2: number analyzed (Participants) | 46 | 0 | 0 | 0
  Month 2 | 4.52 [4.39 to 4.66] |  |  |

2. Primary Outcome: Mean Intervention Appropriateness Measure (IAM) Scale Score
Description: Intervention appropriateness was defined as the perceived relevance and usefulness of the intervention to support decision making about HIV prevention methods. Appropriateness was assessed through self-report using a validated 4-item scale (IAM) to measure women's perceptions of its relevance and usefulness (responses rated on a 5-point Likert scale ranging from 1="Completely Disagree" to 5="Completely Agree"). For each participant at each timepoint, a mean IAM scale score was calculated ranging from 1 to 5. Higher scores indicate greater appropriateness. Individuals' mean IAM scale scores were averaged at each timepoint, and a 95% confidence interval around the mean of means was calculated using the common standard error.
Time Frame: enrollment visit (month 0), month 2 follow up visit
Population: Only participants that received the MyChoice intervention and had one or more completed items of the IAM scale were included. Participants in the Standard of Care (SOC) Control Arm, Male Partner In-Depth Interviews, and Clinician and Counselor In-Depth Interviews were not asked to complete these items.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | My Choice for HIV Prevention (MyChoice) | Standard of Care (SOC) Control Arm | Male Partner In-Depth Interviews | Clinician and Counselor In-Depth Interviews
Number analyzed (Participants) | 50 | 0 | 0 | 0
score on a scale
  Enrollment (Month 0) | 4.59 [4.47 to 4.71] |  |  |
  Month 2: number analyzed (Participants) | 46 | 0 | 0 | 0
  Month 2 | 4.46 [4.32 to 4.61] |  |  |

3. Primary Outcome: Mean Feasibility Intervention Measure (FIM) Scale Score
Description: Intervention feasibility was defined as extent to which the intervention is perceived to be feasible or practical. Feasibility was assessed through self-report using a validated 4-item scale (FIM) to measure women's perceptions of its practicability and ease of use (responses rated on a 5-point Likert scale ranging from 1="Completely Disagree" to 1="Completely Agree"). For each participant at month 0, a mean FIM scale score was calculated ranging from 1 to 5. Higher scores indicate greater feasibility. Individuals' mean FIM scale scores were averaged, and a 95% confidence interval around the mean of means was calculated using the common standard error.
Time Frame: enrollment visit (month 0)
Population: Only participants that received the MyChoice intervention and had one or more completed items of the FIM scale were included. Participants in the Standard of Care (SOC) Control Arm, Male Partner In-Depth Interviews, and Clinician and Counselor In-Depth Interviews were not asked to complete these items.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | My Choice for HIV Prevention (MyChoice) | Standard of Care (SOC) Control Arm | Male Partner In-Depth Interviews | Clinician and Counselor In-Depth Interviews
Number analyzed (Participants) | 50 | 0 | 0 | 0
score on a scale | 4.53 [4.40 to 4.65] |  |  |

4. Secondary Outcome: Mean Decisional Conflict Scale (DCS) Score
Description: A validated scale (DCS) was utilized to assess participants' perceptions decisional conflict regarding the decision whether to use PrEP following receipt of MyChoice or SOC counseling. The 16 items in the scale assess these perceptions by asking participants to rate statements regarding their perceived level of uncertainty, satisfaction, clarity of personal values, and support for decision-making. Responses are rated on a 5-point Likert scale ranging from 0="Strongly agree" to 4="Strongly Disagree". DCS scores range from 0 to 100 points (mean item rating multiplied by 25), with higher scores indicating a higher level of decisional conflict. At month 0 after the intervention, individuals' mean DCS scores were averaged, and a 95% confidence interval around the mean of means was calculated using the common standard error. Only participants that had one or more completed items of the DCS were included.
Time Frame: enrollment visit (month 0)
Population: Participants that received the MyChoice intervention or SOC at month 0 were included if they had at least one non-missing item on the 16-item DCS. Participants in the Male Partner In-Depth Interviews and Clinician and Counselor In-Depth Interviews arms were not asked to complete these items.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | My Choice for HIV Prevention (MyChoice) | Standard of Care (SOC) Control Arm | Male Partner In-Depth Interviews | Clinician and Counselor In-Depth Interviews
Number analyzed (Participants) | 50 | 50 | 0 | 0
score on a scale | 14.8 [10.3 to 19.3] | 18.3 [15.3 to 21.3] |  |
Statistical Analysis 1: Comparison: My Choice for HIV Prevention (MyChoice) vs Standard of Care (SOC) Control Arm; The null hypothesis is that the mean DCS for the MyChoice and SOC arms are equal; Test type: Superiority; p = 0.2157, Welch's t test, 2 sided — The a priori threshold for statistical significance is p<0.05; The Welch's t test statistic was -1.25 and the degrees of freedom were 84.67; Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-8.9 to 1.9], Standard Error of Mean 2.74 — The mean difference was calculated by subtracting the mean DCS of the SOC arm from the mean DCS of the MyChoice intervention arm (MyChoice mean - SOC mean)

ADVERSE EVENTS:
Time Frame: From completion of the baseline visit through the last completed study visit, up to 3 months.
Description: The severity of adverse events (AEs) was graded using the National Institute of Health's Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric AEs.
Arm/Group | My Choice for HIV Prevention (MyChoice) | Standard of Care (SOC) Control Arm | Male Partner In-Depth Interviews | Clinician and Counselor In-Depth Interviews
All-Cause Mortality (participants affected / at risk) | 0/50 | 1/50 | 0/20 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/50 | 0/20 | 0/12
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/20 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | My Choice for HIV Prevention (MyChoice) (N=50) | Standard of Care (SOC) Control Arm (N=50) | Male Partner In-Depth Interviews (N=20) | Clinician and Counselor In-Depth Interviews (N=12)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-02-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT06394323/Prot_001.pdf
  • Statistical Analysis Plan (2025-08-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT06394323/SAP_002.pdf
  • Informed Consent Form (2024-12-09): https://cdn.clinicaltrials.gov/large-docs/23/NCT06394323/ICF_000.pdf